CLINICAL TRIAL: NCT02872740
Title: Gastric Arterial Embolization for Weight Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Martin Simons, BSc, MD, FRCPC, FSIR, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-9576
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Embolization of Left Gastric Artery (Experimental): These patients will have their left gastric artery embolized
  Interventions: Procedure: Embolization of Left Gastric Artery
- Embolization of Gastroepiploic Artery (Experimental): These patients will have their gastroepiploic artery embolized
  Interventions: Procedure: Embolization of Gastroepiploic Artery

INTERVENTIONS:
Procedure: Embolization of Left Gastric Artery — Left gastric artery will be embolized to stasis with 150-250 micron polyvinyl alcohol particles
  Arms: Embolization of Left Gastric Artery
Procedure: Embolization of Gastroepiploic Artery — Gastroepiploic artery will be embolized to stasis with 150-250 micron polyvinyl alcohol particles
  Arms: Embolization of Gastroepiploic Artery

SUMMARY:
Title: Embolization of Gastric Arterial Supply for Weight Loss

Sample size:

10 patients

Study Population: Morbidly obese patients who were seen by the bariatric surgery program at Toronto Western Hospital but are either not interested or not eligible for surgery.

Study Design:

Single center, randomized, prospective, non-blinded pilot study.

Study Duration:

12 months (November 2015 - December 2015).

Agent:

150-250 micron polyvinyl alcohol particles

Primary objective:

To further evaluate the safety of embolization of the left gastric and gastroepiploic arteries. To determine if either or both will result in significant weight loss and decrease in waist circumference among obese patients.

Primary objective measure:

The number of adverse events in a 1 year period will be recorded. The weight change from baseline will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Meet standard eligibility criteria for bariatric surgery. BMI of >= 40 -or- BMI of >=35 with one of the following comorbid conditions: hypertension, type 2 diabetes, obstructive sleep apnea, coronary artery disease

Exclusion Criteria:

Basic

Unable to provide informed consent (legally authorized representative is acceptable) Unable or unwilling to come for follow up appointments Age < 18 or >80 Weight >400 lbs or 180kg due to weight limits on angiographic tables Moderate or severe allergy to iodinated contrast media not amenable to premedication as defined by the ACR contrast guidelines Pregnant, breastfeeding or actively trying to become pregnant in the next year Inability to lie flat for the duration of the procedure Limited life expectancy < 1 year Patient enrolled in another interventional study, they will be permitted to enter this study 30 days after reaching the prior studies primary endpoint Arterial anatomy not feasible for intervention based on investigator assessment

Gastrointestinal

Pre-existing chronic abdominal pain History of inflammatory bowel disease History of gastroparesis Prior history of gastric surgery, embolization or radiation Prior or current history of peptic ulcer disease Significant risk factors for peptic ulcer disease including daily NSAID use, active smoking or active H. Pylori infection Abnormal upper endoscopy Hepatic Cirrhosis Portal venous hypertension Hepatic Bilirubin > 2.0 mg/dL Albumin < 2.5 g/L

Cardiovascular

Known aortic pathology such as aneurysm or dissection Peripheral arterial disease

Renal

Renal insufficiency as evidenced by estimated GFR < 60ml/min.1.73m2

Hematologic/Immunologic/Oncologic/Infectious

Acute or chronic infection Active cancer or prior history of cancer <10 years ago Autoimmune disease requiring immunosuppression Neutrophils < 1.5 x 10^9/L Platelets < 50 x 10^9/L INR >1.7

Psychiatric

Major diagnosed psychiatric comorbidities such a major depressive disorder, schizophrenia, bipolar disorder that are deemed to likely interfere with follow up History of an eating disorder such as anorexia or bulimia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 1 year
  Adverse events

SECONDARY OUTCOMES:
Weight | 1 year
  weight change
Cardiovascular risk factors | 1 year
  serum lipids, hemoglobin A1C, blood pressure, sleep apnea

IPD SHARING:
Plan to Share IPD: No